CLINICAL TRIAL: NCT06097221
Title: The Advance Project - Advancing Sleep Timing to Improve Depression, a Randomised Clinical Trial.
Brief Title: The Advance Project - Advancing Sleep Timing to Improve Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Klaus Martiny, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADVANCE
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Advance-group (Experimental): The group will recieve 8 hours of psychotherapy with focus on advancing sleep timing, besides their treatment as usual.
  Interventions: Behavioral: CRT-Advance
- Control-group (Active Comparator): Treatment as usual at the outpaitent unit.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: CRT-Advance — Psychotherapy with focus on advancing sleep timing, using diaries on sleep and zeitgebers.
  Arms: Advance-group
Behavioral: Treatment as usual — Treatment as usual in the outpatient psychiatric unit.
  Arms: Control-group

SUMMARY:
150 patients with moderate to severe depression, recently discharged from a psychiatric ward and now recieving treatment at an outpatient unit at Mental Health Center Copenhagen, will be randomised in to two groups. A treatment ad usual (TAU) group and an Advance-group. The Advance-group will receive a psychotherapeutic intervention focusing on advancing sleep timing to improve depression.

DETAILED DESCRIPTION:
Objective Patients treated at outpatient psychiatric services for major depression improves slowly from their depression despite use of psychopharmacological, psychological, and supportive methods. This is in many cases due to severe sleep disturbances as part of their current depressive episode. Typically, these patients have difficulties keeping their habitual sleep-wake cycle, that drifts to later in the evening and morning. Thus, patients who, before being depressed, sleeps around 11 PM and wake up around 7 AM, often drift to a later sleep schedule at around 1 AM and a wake-up time at 9 AM or even later during their depressive period. The reason for the drift of the sleep schedule is mainly caused by reduced signals to the circadian system from daylight, social input, dieting and exercise. This reduced input is partly a result of the changed behavior of patients due to their depressive symptoms making them less structured, less socially active, less physically active, eating erratically, and staying more indoors thereby receiving less daylight. Another reason for the sleep drift is the presence of diurnal variation of depressive symptoms with morning worsening and evening improvement tempting patients to stay up later because of the better evening mood. The sleep drift makes patients out of synchrony with societal and workplace rhythms, and the investigators have clinical and research evidence for mood worsening associated with sleep drift and of improvement of depression when patients correct their sleep drift.

The physiological background behind why late sleep worsens and maintain depression is thought to be caused by a sleep induced inhibition of the raphe nuclei in the brain stem downregulating the serotonergic activity in the forebrain in the late phase of the sleep period.

The association between depression and sleep/sleep timing is well established from the bulk of literature on sleep deprivation, and sleep phase advance. Regulation of sleep disturbances thus has a great potential as a specific new treatment target.

Our recent study showed that a newly developed psychoeducation method, Circadian Reinforcement Therapy (CRT) could prevent sleep drift and improve mood in patients discharged from inpatient wards. The standard psychoeducation manuals used at psychiatric services do not focus adequately on the relation between signals to the circadian system, sleep timing, and mood. The principle in the CRT is based on scientific findings that sleep timing and thus mood is for a large part a result of how the actual day is spend - what signals is reaching the circadian system. The influence of light during the day is termed Prior Light History and has been documented to influence sleep, circadian rhythms, and melatonin secretion/suppression. The main time signals to the circadian system (zeitgebers) are light (electrical or daylight), social activity, exercise, and diet. The CRT method aimed to strengthen all these time signals and normalize the sleep timing leading to improvement of depression.

The objective of this project is to investigate whether the use of an adjusted CRT method named CRT-Advance focusing even more on advancement of the sleep-wake cycle can induce an antidepressant effect in selected patients that have drifted in their sleep during their depressive episode (enriched sample).

The Advance method acknowledges the importance of clinical contact between project staff and patients. In addition, patients will be asked to wear activity watches that measures light exposure and sleep/wake timing. Tracking participants individual behavior by accelerometers helps to reveal the invisible timing of the circadian system.

If the CRT-Advance method is effective, it can be established on a wider scale in psychoeducation manuals and guidelines for depression and the method can have a potential for psychiatric services making their treatment more cost-effective. An important point is that traditional treatment methods such as pharmacotherapy and psychotherapy is less effective in the presence of significant sleep problems due to daytime sleepiness and the depressiogenic effect of mistimed sleep.

On a societal scale, there is a large need for treatments for insomnia, and the investigators also expect the CRT-Advance method to improve insomnia by reducing sleep onset problems through the advancement of sleep timing. This could reduce the use of dependence inducing hypnotics.

The number of non-pharmacological treatment methods are now growing as psychotropic drugs often are often associated with severe side effects and often a lack of efficacy. Therefore, there is a need for the testing of novel treatment methods based on existing theoretical background.

Chronotherapy has provided evidence based new treatment options like light therapy, wake therapy, sleep time stabilization, and lately dark therapy. The chronotherapeutic research field consists of a growing number of international research groups and societies, largely interdisciplinary, with basic researchers and clinicians around the world.

The investigators also see a steady growth in the interest of chronotherapeutic application in Denmark (https://psy.au.dk/en/circadianpsychology).

With several new professorships in the field, this proposed project is highly likely to inspire the field further, making it easier to attract funding for research positions and international collaboration.

Methods The design is a randomised clinical trial (RCT), where participants with major depression and delayed sleep timing will be randomised into either a treatment as usual (TAU) group or a CRT-Advance group using psychoeducation methods to reset sleep timing to earlier. The CRT-Advance method is based on the use of (1) sleep diaries, (2) zeitgebers diaries diaries capturing time signals to the circadian system e.g. daylight, social contact, meals, and exercise), (3) close clinical weekly contact with focus on the result on sleep and mood of the psychoeducative method.

Actigraphy is recorded with the MotionWatch 8 (MW8, Camntech, UK), which provides an objective measure of sleep timing, 24-hour activity, night-sleep duration, night awakenings, sleep efficiency, day-time napping, and light exposure. Its algorithms on sleep have been validated against polysomnography.

The MW8 is a wristwatch-like device that monitors activity levels and light levels for continuous periods, using accelerometer and light sensing technology. Specialised software (MotionWare Software) analyses data on sleep and circadian activity. Data can be directly downloaded from the watch using a simple USB cable. The MotionWatch 8 will be handed over at inclusion with detailed instructions. During the recording period, the participants will be encouraged to wear the watch continuously day and night. Patients are informed to use the marker button on the device to indicate when they intent to go to sleep (puts away book/phone/etc. and turns off lights). The investigator will download data at each study visit.

Psychoeducation material will be provided individually as part of the weekly clinical contact.

Patients will be followed weekly for eight weeks, thus each patient will receive nine sessions during the project - first visit on day 0, here after one visit every week for eight weeks. The patients must show up at the outpatient treatment unit for the sessions at day 0, week 2, week 4, week 6 and week 8 (final visit). The sessions at week 1, week 3, week 5 and week 7 will be offered as physical meetings as well but can be done over the phone if this is better for the patient.

The primary outcome is change in Hamilton Depression rating scale (HAM-D6) scores from baseline to endpoint (self-rating).

Secondary outcomes are changes in sleep-midpoint, sleep onset and wake-up time from baseline to endpoint from the sleep diaries and based on activity tracking with the MotionWatch 8.

Exploratory outcomes are scores change from baseline to endpoint on the following questionnaires:, Pittsburgh Sleep Quality Index (PSQI, self-rating), WHO Five Well Being Index (WHO-5, self-rating), Insomnia Severity Index (ISI, self-rating), Dysfunctional Believes and Attitudes about Sleep (DBAS, self-rating), Epworth Sleepiness Scale (ESS, self-rating) and Morningness-Eveningness Questionnaire (MEQ, self-rating). Furthermore, the investigators will describe light exposure in the two groups. The sensors will be able to discern when patients are in daylight. The investigators will also describe results from the sleep diaries and the chrono-schedule.

All patients will use the Motion Watch 8 for implementing and validating changes of sleep timing. Adverse events will be monitored. The project will follow GCP regulations and will be approved by the Ethical Committees and the Danish Data Protection Agency.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to major depression (DSM-V)
* Discharge from psychiatric ward within last 30 days
* Sleep onset and/or sleep off-set delayed minimum 1 hour based on the last three days, comparred to sleep in the last week of admittance at the psychiatric ward.

Exclusion Criteria:

* Psychotic depression.
* Cognitive problems making participation difficult.
* Substance abuse (e.g. alcohol).
* Increased suicidal risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | at inclusion, at two weeks, at fourweeks, at six weeks, and at endpoint (after eight weeks)
  Patients will do af self-rating with the Beck Depression IInventory-II self-rating scale. Minimum score is 0, maximum score is 63. A higher score indicates a worsening of depression symptoms

SECONDARY OUTCOMES:
Changes in sleep-midpoint | At inclusion and at endpoint (after eight weeks)
  Measured both with sleep diaries and with actigraphy
Changes in time for sleep onset | At inclusion and at endpoint (after eight weeks)
  Measured both with sleep diaries and with actigraphy
Changes in time for sleep wake-up | At inclusion and at endpoint (after eight weeks)
  Measured both with sleep diaries and with actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny, Professor, Study Director — Mental Health Center Copenhagen
Locations (1):
- Mental Health Center Copenhagen, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No